CLINICAL TRIAL: NCT02841852
Title: Inappropriate Prescribing of Proton-pump Inhibitor is it Associated With the Burden of Comorbidities in Older Patients Over 75 Years Old ?
Brief Title: Inappropriate Prescribing of Proton-pump Inhibitor is it Associated With the Burden of Comorbidities in Older Patients?
Acronym: IPP SA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC13_0262
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Geriatric Disorder

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Proton pump inhibitors (PPIs) are one of the most frequently prescribed classes of drugs in the world and the most effective drugs available to reduce gastric acid secretion. However, studies have shown that PPIs are not always prescribed with a clear indication. Indeed, between 25% and 86% of older individuals taking a PPI have been overprescribed these medications. In older patients, overprescribing of a PPI is associated with increases in morbidity, adverse drug events, hospitalization, and mortality. The hypothesis is that overprescription of PPIs is associated with the individual multimorbidities in older patients evaluated using the multimorbidities group criteria included in the CIRS. The aim of the present study was to establish a relationship between overprescribing of PPIs and multimorbidities in older patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 75 years or more
* Patients hospitalized in geriatric short stay
* Patients with an inhibitor therapy proton pump short geriatric entry
* Patients who have given their written consent

Exclusion Criteria:

* Patients who have expressed their inability or refusal to sign an informed consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients aged 75 and over hospitalized in acute geriatric medicine
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Burden of comorbidities | 48 hours after the entry into acute geriatric medicine
  Burden of comorbidities is assessed by the CIRS (Cumulative Illness Rating Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Laure De DECKER, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Centre Hospitalier de St Nazaire, Saint-Nazaire, France

IPD SHARING:
Plan to Share IPD: Undecided